CLINICAL TRIAL: NCT02485171
Title: Post-fall Syndrome of the Aged Person : Contribution of SAFEWALKER for Rehabilitation
Brief Title: SAFEWALKER Contribution to the Rehabilitation of Older People After a Post-fall Syndrome
Acronym: SAFEER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Safe Step and Walk Movement (SSWM), Toulouse, France (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC31/14/7420
Record Dates: First submitted 2015-06-11; First posted 2015-06-30 (Estimated); Last update posted 2025-12-10 (Actual); Status verified 2018-05

CONDITIONS: Post-fall Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Experimental): Introduction of a walking aid device SAFEWALKER for elderly patients during rehabilitation after a post-fall syndrome.
  Interventions: Device: SAFEWALKER
- No intervention (No Intervention): No introduction of a walking aid device for elderly patients during rehabilitation after a post-fall syndrome.

INTERVENTIONS:
Device: SAFEWALKER — Medical device walking aids.
  Arms: Experimental

SUMMARY:
The main objective of this study is to evaluate the feasibility and acceptability of the use of the robot "SAFEWALKER" complement classical rehabilitation in a group of elderly patients over 70 years during the rehabilitation of post-fall syndrome.

DETAILED DESCRIPTION:
The post-fall syndrome is an acute functional complications of falls that affects nearly one in five elderly fallers. It combines phobia of the previous vacuum, axial and hypertension astasia abasia.

Unrecognized and untreated, it progresses to a major regressive syndrome, severe physical, psychological and social implications. Only an early rehabilitation for an early resumption of walking, prevents such a development.

The main element is to support and encourage the subject to walking. In practice, it was found that the physiotherapist can not be present daily and the duration of its intervention is often short-lived.

This study will examine the contribution of a medical device of a walking aid (SAFEWALKER the robot) in the rehabilitation and empowerment of seniors with a post-fall syndrome. The SAFEWALKER, which is a walking aid device (http://www.safewalker.com), completes the support action exercised by a third person, by reducing support and securing travel. It allows the subject to move alone at will and is a continuity in relation to the management of the physiotherapist, a potential source of motivation.

The hypothesis is that the SAFEWALKER device can be complementary to the walking rehabilitation in post-fall syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized for the treatment of post-fall syndrome

Exclusion Criteria:

* Demential pathology (Mini Mental State <20)
* Parkinson's disease and other degenerative neurological disorders
* Stroke sequelae
* Fractures members in the previous 12 months
* Lower limb prostheses in place within 6 months prior
* Psychiatric disease
* Presence of mucocutaneous lesions perineal
* Obesity (weight >120 kg)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-06-10 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of Safewalker | Day 14
  Number of steps performed at each of the rehabilitation sessions A composite measure based on questionnaires assessing the feasibility (patient and therapist).
Acceptability of Safewalker | Day 14
  A composite measure based on questionnaires assessing the acceptability (patient and therapist).

SECONDARY OUTCOMES:
Walking speed | Day 14
  This parameter will be collected by a pedometer (manual and electronic) and embedded soles (Dynafoot ®) and motion sensors (Bioval ®).
Retropulsion degree | Day 14
  This parameter will be collected by a pedometer (manual and electronic) and embedded soles (Dynafoot ®) and motion sensors (Bioval ®).
Step length | Day 14
  This parameter will be collected by a pedometer (manual and electronic) and embedded soles (Dynafoot ®) and motion sensors (Bioval ®).
Number of falls during the study | Day 14
  The nurse will report the number of times that the patient fell during his hospitalization
Quality of life | Day 14
  Using the Short Form 36 scale
Independence in basic activities of daily living | Day 14
  Using the Activities of Daily Living scale
The fear of falling | Day 14
  Using the Falls Efficacy Scale International

CONTACTS AND LOCATIONS:
Overall Officials: Fatemeh NOURHASHEMI, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Nourhashemi Fatemeh, Toulouse, MIDI Pyrenees, France

REFERENCES:
- [Result] Piau A, Krams T, Voisin T, Lepage B, Nourhashemi F. Use of a robotic walking aid in rehabilitation to reduce fear of falling is feasible and acceptable from the end user's perspective: A randomised comparative study. Maturitas. 2019 Feb;120:40-46. doi: 10.1016/j.maturitas.2018.11.008. Epub 2018 Nov 17. PMID 30583763